CLINICAL TRIAL: NCT03660891
Title: Observational Study Measuring Neuromuscular Block Depth by a TOF or PTC Monitor on the Thumb and on the Upper Arm of the Same Side.
Brief Title: OS NMB Depth Measured by Central and Peripheral Monitor.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jan Mulier, principle investigator, AZ Sint-Jan AV
Other Study IDs: OS NMBcentralperipheral
Record Dates: First submitted 2018-08-19; First posted 2018-09-07 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: measuring neuromuscular block — During anesthesia patients are monitored with two instead of one NMT monitor. the difference in measured TOF-PTC is compared

SUMMARY:
Comparing during anesthesia in the same patient 2 neuromuscular monitors on the same arm.

DETAILED DESCRIPTION:
NMT (neuromuscular transmission) depth can be measured at the same arm with two different methods during clinical practice.

the first (TOF Watch) measures the musculus adductor pollicis acceleration while the second method (TOF Cuff Monitor) uses a blood pressure cuff to measure the pressure changes induced by the upper arm muscles.

During general anesthesia when NMB (neuromuscular block) is required both methods are used. Every 5 minutes, if clinical required, the NMB is monitored by TOF-PTC. If the measurement of TOF is zero the monitor continues by measuring PTC ( the system will measure TOF followed by PTC if TOF is zero) TOF-PTC is recorded and later compared for identity or systematic difference in one or the other direction.

The measured answer can be TOF 4 (4 answers) with a ratio between answer 1 and 4 expressed and a percentage, TOF 3 (3 answers), TOF 2, TOF 1, TOF 0 + PTC 20, TOF 0 + PTC 19, up to TOF 0 + PTC 0

ELIGIBILITY:
Inclusion Criteria: all patients scheduled for an elective surgery requiring neuromuscular block during anesthesia

* laparoscopic surgery of upper abdomen including all types of bariatric surgery.

Exclusion Criteria: not possible to measure NMT (neuromuscular transmission) by cuff or thumb monitor

* upper arm obesity excluding the use of an upper arm blood pressure cuff
* allergy to NMB (neuromuscular blockers)
* contra indication for a deep NMB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients undergo a laparoscopic surgery and require a deep NMB.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
TOF-PTC value | From induction of anesthesia (intubation with ETT) till end of anesthesia (extubation of ETT) most frequent between 1 and 2 hours, max 6 hours in duration
  Difference in TOF-PTC measured by two different devices during anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Paul Mulier, Principal Investigator — AZSint Jan AV
Locations (1):
- Azsintjan, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No